CLINICAL TRIAL: NCT01940562
Title: Eltrombopag for Enhancing Platelet Engraftment in Pediatric Patients Undergoing Cord Blood Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: moshe yeshurun (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, moshe yeshurun, Head, BMT unit, Rabin Medical Center, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0195-13
Record Dates: First submitted 2013-09-08; First posted 2013-09-12 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Pediatric Patients Undergoing Allogeneic Cord Blood Transplantation.
Keywords: cord blood transplantation; platelets; eltrombopag
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Pediatric patients undergoing allogeneic UCB transplantation will receive eltrombopag from day +1 until platelet count has exceeded 50,000/microliter for 14 consecutive days without platelet transfusion.
  Starting doses are 100 mg/d for children >40 kg body weight (BW), 50 mg/d for children 20-40 kg BW, and 2 mg/kg/d for children <20 kg BW.
  If unsupported platelet count has not reached the threshold of 20,000/microliter, doses will be escalated every 2 weeks up to maximal doses of 200 mg/d for children ≥ 40 kg BW, 150 mg/d for children 20-40 kg BW and 3.5 mg/kg for children <20 kg BW.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — Children ≥= 40 kg BW:
  From day +1, start eltrombopag 100 mg/d. If primary end point not reached on day +14, then from day +15 - 150 mg/d. If primary end point not reached on day +28 then from day +29 - 200 mg/d (maximal dose).
  Children 20-40 kg BW:
  From day +1, start eltrombopag 50 mg/d. If primary end point not reached on day +14, then from day +15 - 75 mg/d. If primary end point not reached on day +28 then from day +29 - 100 mg/d.If primary end point not reached on day +42, then from day +43 and on - 150 mg/d (maximal dose).
  Children < 20 kg BW:
  From day +1, start eltrombopag - 2 mg/kg/d. If primary end point not reached on day +14, then from day +15 - 3 mg/kg/d. If primary end point not reached on day +28 then from day +29 - 3.5 mg/kg (maximal dose).
  If present dose not tolerated, return to last tolerated dose. Eltrombopag will be discontinued after platelet count has exceeded 50,000/microliter for 14 consecutive days without administration of platelets.
  Other Names: Revolade

SUMMARY:
Platelet recovery is significantly hampered following umbilical cord blood transplantation (UCB). Thus, after UCB transplantations, patients are platelet transfusion-dependent for prolong periods of time.

Eltrombopag is a thrombopoietin-receptor agonist that initiates thrombopoietin-receptor signaling and thereby induces proliferation and maturation of megakaryocytes.

We will evaluate the safety and efficacy of eltrombopag for enhancing platelet engraftment in pediatric patients undergoing cord blood transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 1 year and < 18 years old.
2. Patients receiving unmanipulated single or double UCB allogeneic grafts.
3. Malignant and non malignant indications for transplantation.
4. Myeloablative and reduced intensity conditioning regimens.
5. Patients must meet all other pre-transplantation criteria of the transplantation center including acceptable tests of heart, liver, kidney, and lung function (standard screening for transplantation per PI, and co-investigators).
6. Written informed must be obtained from the patient's guardian, and accompanying informed assent from the patient for children over 6 years old.
7. Able to comply with study protocol.

Exclusion Criteria:

1. Indications for transplantation

   1. Patients with primary myelofibrosis.
   2. French-American-British classification (FAB)M7 acute myeloid leukemia. Acute leukemia secondary to a myeloproliferative neoplasm.
   3. Patients with persistent acute leukemia (>5% bone marrow blasts) at the time of transplantation.
2. Patients with prior thromboembolic event. Patients with previous catheter related thrombosis will be eligible if more than 3 months elapsed.
3. Hypersensitivity to eltrombopag.
4. Liver enzymes abnormalities:

Alanine aminotransferase (ALT) levels > 3 times the upper limit of normal (ULN) or serum bilirubin > 1.5 ULN (unless due to Gilbert's syndrome or hemolytic bilirubin).

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Platelet engraftment rate up to 50 days post transplantation, defined as the first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter. | 50 days

SECONDARY OUTCOMES:
Time to partial platelet engraftment, defined as the first of 7 consecutive days of an unsupported platelet count of at least 20,000/microliter. | 180 days
Time to sustained complete platelet engraftment defined as the first of 7 consecutive days of an unsupported platelet count of at least 50,000/microliter. | 180 days
Complete platelet engraftment rates up to 50 days post transplantation defined as the first of 7 consecutive days of an unsupported platelet count of at least 50,000/microliter. | 50 days
Time to neutrophil engraftment defined as the first of 3 consecutive days to achieve an absolute neutrophil count ≥ 500/microliter. | 60 days

OTHER OUTCOMES:
Any grade 3/4 adverse event | 12 months
  Number of participants with any grade 3/4 adverse event as a measure of safety and tolerability.
Thromboembolic events | 12 months
  Number of participants with a thromboembolic event as a measure of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Yeshurun, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Hadassah hospital, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva